CLINICAL TRIAL: NCT06261320
Title: Mesotherapy Treatment of Irritable Bowel Syndrome
Acronym: MESOCOLO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Polyclinique de l'Europe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506950-18-00
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: mesotherapy; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesotherapy; Trimecaine; thiocolchicoside; Amitriptyline; Pyrrolidonecarboxylic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Mesotherapy with mesocaine, thiocolchicoside, amitriptyline, magnesium pidolate

INTERVENTIONS:
Drug: Mesotherapy with mesocaine, thiocolchicoside, amitriptyline, magnesium pidolate — 4 sessions of mesotherapy (mesocaine, thiocolchicoside, amitriptyline, magnesium pidolate), with intra-epidermal and intra-hypodermal technics.

SUMMARY:
Irritable bowel syndrome (IBS) is a gastrointestinal transit disorder characterized by chronic abdominal pain and impaired transit in the absence of demonstrated organic disease. Considered a non-fatal disease, its effects relate more to quality of life, work production and health care systems.

Given the complexity of this disease, no treatment has been recognized as standard treatment. The treatment is rather focused on treating the symptoms caused (chronic pain or intestinal transit disorder). In general, therapy is considered individualized and includes lifestyle/diet modifications and pharmaceutical therapy.

Several published case studies evaluating the effect of mesotherapy on improving the severity of the disease have demonstrated an improvement in the symptoms of this syndrome. Due to the limited number of case studies and the insufficient level of evidence to conclude, our study will therefore be a before-and-after intervention study, to evaluate the effect of four mesotherapy sessions on the treatment of IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from Irritable Bowel Syndrome according to the Rome IV criteria, whose diagnosis was made by a specialist in Hepato-Gastro-Enterology,
* Francis score >75/500, i.e. minimal, moderate or severe severity,
* Patient who has failed conventional treatment (treatment followed for at least 1 year and not showing an improvement in symptoms)
* Absence of risk of ongoing pregnancy in women of childbearing age, validated by a urine test during the first consultation and before treatment and each month during treatment and until 1 month after the end of treatment

Exclusion Criteria:

* Patient with the following medical history or current pathologies: organic gastrointestinal pathology, disabling neurological pathology, disabling psychiatric pathology
* Recent Post Traumatic Stress Syndrome (<1 year),
* Fibromyalgia syndrome,
* Known allergy to medications used in mesotherapy treatment,
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale(IBS-SSS) | day 8, day 15, day 30, day 45
  Includes 5 items regarding pain (intensity and number of days), abdominal distention, satisfaction of bowel habit, and interference of daily life of the last 10 d on a 10-point scale.
  Gives a score between 0 and 500, and groups of severity can be made: mild (≤175), moderate (175-300), and severe (≥300) IBS.

SECONDARY OUTCOMES:
Functional Digestive Disorders Quality of Life questionnaire (FDDQL) | day 30, day 45
  43 items with 8 subscales : daily activity, anxiety, nutrition, sleep, discomfort, health perception, adaptation and impact of stress Global score is between 0 and 100.
Pain evaluation | day 8, day 15, day 30, day 45
  Evaluation of pain with a scale from 0 (no pain) to 10 (worst pain imagined)
Global satisfaction | day 45
  4 questions with Likert scale of 5 items, to "not at all satisfied" to "very satisfied"
Anxiety evaluation : Questionnaire "Hospital anxiety and depression scale" | day 30, day 45
  14 items with 7 about depression and 7 about anxiety. Each item is noted with a Likert scale of 4 points, from 0 (no symptoms) to 3 (strong symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique de l'Europe, Saint-Nazaire, France

IPD SHARING:
Plan to Share IPD: No